CLINICAL TRIAL: NCT00566150
Title: Levetiracetam in the Management of Bipolar Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0508000506
Record Dates: First submitted 2007-11-29; First posted 2007-12-03 (Estimated); Results first posted 2015-11-02 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2016-08

CONDITIONS: Bipolar Depression
Keywords: Keppra; Levetiracetam; Anticonvulsant; Depression; Bipolar Disorder; Affective Disorders; Mood Disorders; Double Blind; Acute Antidepressant Effects
MeSH Terms: conditions — Bipolar Disorder; Depression; Mood Disorders | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levetiracetam (Active Comparator)
  Interventions: Drug: Levetiracetam
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levetiracetam — Flexible dose up to 2500mg per day, for 6 weeks.
  Other Names: Keppra
  Arms: Levetiracetam
Drug: Placebo — Flexible dose up to 2500mg per day, for 6 weeks.
  Arms: Placebo

SUMMARY:
A 6-week outpatient, double-blind, placebo-controlled, add-on trial to investigate the effects of levetiracetam on depressive symptoms in bipolar depressed patients.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of bipolar disorder
* Presence of a current major depressive episode on the SCID
* Score of 17 or great on the HDRS
* Capable of giving voluntary written consent

Exclusion Criteria:

* Significant current substance dependence/abuse within 3 months preceding the trial
* Active suicidal ideation
* Pregnant/lactating mothers
* Significant medical history

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-10; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zubin Bhagwagar, MD PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Background] Muralidharan A, Bhagwagar Z. Potential of levetiracetam in mood disorders: a preliminary review. CNS Drugs. 2006;20(12):969-79. doi: 10.2165/00023210-200620120-00002. PMID 17140277
- [Derived] Saricicek A, Maloney K, Muralidharan A, Ruf B, Blumberg HP, Sanacora G, Lorberg B, Pittman B, Bhagwagar Z. Levetiracetam in the management of bipolar depression: a randomized, double-blind, placebo-controlled trial. J Clin Psychiatry. 2011 Jun;72(6):744-50. doi: 10.4088/JCP.09m05659gre. Epub 2010 Oct 19. PMID 21034692

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 2005-2008 from New Haven, CT and surrounding areas.
Groups:
- Levetiracetam: Subjects on active study medication.
- Placebo: Subjects assigned to placebo control group.
Period: Overall Study
Arm/Group | Levetiracetam | Placebo
Started | 19 | 16
Completed | 10 | 11
Not Completed | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levetiracetam | Placebo | Total
Number analyzed (Participants) | 19 | 16 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 16 | 35
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (10.7) | 42.4 (9.6) | 44.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 19 | 16 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Depression Rating Scale (HDRS-21) Total Score From Baseline at Week 6.
Description: Change is observed value at each visit minus baseline value. HDRS-21 is a 21-item instrument measuring depression. Items are rated on a scale from 0 (symptoms not present) to a maximum of 2 to 4 (symptom extremely severe) for a total score range of 0 to 60.
Time Frame: Baseline to week 6
Population: Weeks 1-6 are Intent to treat (ITT) population Observed Cases. All participants included received at least 1 dose of study intervention and at least 1 assessment post-baseline.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Levetiracetam | Placebo
Number analyzed (Participants) | 17 | 15
score on scale
  Week 1 (n=17, n=15) | -2.7647 (1.4138) | -4 (1.5051)
  Week 2 (n=15, n=14) | -3.4259 (1.4618) | -6.5875 (1.5327)
  Week 3 (n=13, n=14) | -2.1243 (1.5441) | -6.3625 (1.5458)
  Week 4 (n=11, n=13) | -4.3534 (1.6582) | -6.3851 (1.583)
  Week 5 (n=11, n=13) | -6.952 (1.7105) | -6.4368 (1.6006)
  Week 6 (n=10, n=11) | -4.8136 (1.7806) | -7.0712 (1.6838)
Statistical Analysis 1: Comparison: Levetiracetam vs Placebo; Comparison of changes in outcome between treatment groups at week 6; Test type: Superiority or Other; p = 0.29, Mixed Models Analysis — Unadjusted. Statistical significance was p<0.05; Fixed categorical effects: group (as a between-subjects factor), time (as a within-subjects factor), group x time interaction

2. Secondary Outcome: Change in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score From Baseline at Week 6.
Description: Change is observed value at each visit minus baseline value. MADRS is a 10-item instrument measuring depression: scale range between 0(normal) - 6(most abnormal)for each item. Total possible score is 0 - 60.
Time Frame: Baseline to week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Levetiracetam | Placebo
Number analyzed (Participants) | 17 | 15
score on scale
  Week 1 (n=17, n=15) | -3.2941 (2.0145) | -2.7333 (2.1446)
  Week 2 (n=15, n=14) | -5.2319 (2.1105) | -7.256 (2.1999)
  Week 3 (n=13, n=14) | -3.384 (2.2162) | -9.0417 (2.1999)
  Week 4 (n=11, n=13) | -5.5505 (2.3441) | -8.7608 (2.2514)
  Week 5 (n=11, n=12) | -9.9142 (2.3441) | -6.6591 (2.3061)
  Week 6 (n=10, n=11) | -6.5208 (2.4183) | -4.5153 (2.3691)
Statistical Analysis 1: Comparison: Levetiracetam vs Placebo; Comparison of changes in outcome between treatment groups at week 6; Test type: Superiority or Other; p = 0.07, Mixed Models Analysis — Unadjusted. Statistical significance was p<0.05; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Subjects Who Achieve Remission.
Description: Remission response is measured as an HDRS-21 total score is less than or equal to 7.
  HDRS-21 measures range of depressive symptoms. Endpoint is LOCF.
Time Frame: Week 6
Measure: Number; unit: Participants
Arm/Group | Levetiracetam | Placebo
Number analyzed (Participants) | 17 | 15
Participants
  Remitted | 0 | 4
  Not remitted | 17 | 11
Statistical Analysis 1: Comparison: Levetiracetam vs Placebo; Week 6; Test type: Superiority or Other; p = .038, Fisher Exact — Statistical significance was p<0.05; Fisher's exact test was used to test for significance between groups

4. Secondary Outcome: Change in Clinical Global Impressions Scale for Bipolar Disorder (CGI-BP) Depression Severity Rating From Baseline at Week 6.
Description: Change is observed value at each visit minus baseline value. CGI-BP depression severity is an instrument which measures severity of depression in bipolar disorder. Scale range: 1=normal, not ill; 7=very severely ill
Time Frame: Baseline to week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Levetiracetam | Placebo
Number analyzed (Participants) | 17 | 15
score on scale
  Week 1 (n=17, n=15) | -0.2941 (0.1982) | -0.4667 (0.211)
  Week 2 (n=14, n=14) | -0.3186 (0.211) | -0.6956 (0.2161)
  Week 3 (n=13, n=14) | -0.1984 (0.2207) | -0.7753 (0.2177)
  Week 4 (n=11, n=13) | -0.3729 (0.2386) | -0.8403 (0.2238)
  Week 5 (n=11, n=12) | -0.7325 (0.244) | -0.8739 (0.2322)
  Week 6 (n=10, n=10) | -0.5742 (0.2539) | -0.9294 (0.2505)
Statistical Analysis 1: Comparison: Levetiracetam vs Placebo; Comparison of changes in outcome between treatment groups; Test type: Superiority or Other; p = 0.79, Mixed Models Analysis — Unadjusted. Statistical significance was p<0.05; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected during course of the study and for two weeks after last study intervention.
Arm/Group | Levetiracetam | Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/16
Other Adverse Events (participants affected / at risk) | 17/19 | 15/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Levetiracetam (N=19) | Placebo (N=16)
Somnolence (Nervous system disorders) | 10 | 7
GI symptoms (Gastrointestinal disorders) | 6 | 5
Irritability (Psychiatric disorders) | 5 | 1
Coordination (Nervous system disorders) | 4 | 0
Shakiness (Nervous system disorders) | 2 | 2
Dizziness (Nervous system disorders) | 3 | 2
Weakness (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 3 | 6
Dry mouth (Gastrointestinal disorders) | 2 | 2
Hypomanic symptoms (Psychiatric disorders) | 2 | 0
Worsening of depressive symptoms (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Slurred speech (Nervous system disorders) | 1 | 0
Sunstance Abuse Relapse (Psychiatric disorders) | 2 | 1
Increase in suicidality (Psychiatric disorders) | 1 | 0
Cognitive (Psychiatric disorders) | 1 | 1
Drooling (Gastrointestinal disorders) | 1 | 0
Genitourinary (General disorders) | 1 | 0
Blurred vision (Nervous system disorders) | 0 | 1
Unusual dreams/nightmares (General disorders) | 0 | 1
Taste (Gastrointestinal disorders) | 0 | 1
Nosebleed (General disorders) | 0 | 1
Cardiac (Cardiac disorders) | 0 | 1
Rash (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle soreness (Musculoskeletal and connective tissue disorders) | 0 | 1
Cold (General disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No